CLINICAL TRIAL: NCT03940625
Title: Anthracycline Induced Cardiotoxicity - Early Detection by Combination of Diastolic Strain and T2-mapping
Acronym: ANKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-002
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Myocardial Damage; Cardiotoxicity
Keywords: breast cancer; antracyclines; cardiotoxity; myocardial damage; MRI; T2 mapping; diastolic function; echocardiography; early detection; strain analysis
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI and echocardiography, laboratory parameters — Cardiac MRI including cine imaging (volumetric determination of LV-EF), late gadolinium enhancement, strain analysis, T1 mapping and T2 mapping Echocardiography including 3D-EF, diastolic function and strain analysis Determination of laboratory parameters including cardiac enzymes (Troponin T and high sensitivity Troponin T) and cardiac markers (BNP and NT-pro BNP)

SUMMARY:
Anthracyclines (e.g. Doxorubicin) are an important and highly effective chemotherapeutic. They are used in various tumor entities and are established for breast cancer treatment. The most significant prognostic side effect is cardiotoxicity, which occurs in up to 50 patients. Female gender must be considered an independent risk factor for the incidence and severity of associated heart failure. The aim of this study is to demonstrate that dose-dependent anthracycline-induced cardiotoxicity has a measurable effect on T2 mapping on MRI. The second aim is to demonstrate if the combination of diastolic strain (echo and MRI) and T2 mapping can detect earlier anthracycline-induced myocardial damage than via the established method of the echocardiographic measurement of LV-EF and the conventional quantification of diastolic function.

DETAILED DESCRIPTION:
In order to answer the question, patients with breast cancer, who will undergo a chemotherapeutic treatment with antracycline, will be examined before chemotherapy (including cmr and echocardiography) and after chemotherapy at different times within one year.

ELIGIBILITY:
Inclusion Criteria:

* Planned therapy with an anthracycline and at least 1 year follow up
* >18 years of age
* written informed consent

Exclusion Criteria:

* prior cardiovascular disease
* diabetes mellitus
* previous therapy with anthracyclines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
reduction of the left ventricular ejection fraction (LV-EF) by 10% to under 50% | after 12 months
  volumetric determination of LV-EF

SECONDARY OUTCOMES:
reduction of the left ventricular global longitudinal strain (GLS) by over 15% | after 12 months
  determination of GLS via strain analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Voss F, Nienhaus F, Pietrucha S, Ruckhaberle E, Fehm T, Melz T, Cramer M, Haberkorn SM, Flogel U, Westenfeld R, Scheiber D, Jung C, Kelm M, Polzin A, Bonner F. Anthracycline therapy induces an early decline of cardiac contractility in low-risk patients with breast cancer. Cardiooncology. 2024 Jul 16;10(1):43. doi: 10.1186/s40959-024-00244-y. PMID 39014463